CLINICAL TRIAL: NCT03868800
Title: Shared Decision-Making and Dialysis Choice: A Complex Intervention
Brief Title: Shared Decision-Making and Dialysis Choice
Acronym: SDM-DC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Hillerod Hospital, Denmark (Other); Hospital of Southern Jutland (Other); Regional Hospital Holstebro (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 04032019
Record Dates: First submitted 2019-03-07; First posted 2019-03-11 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SDM-DC (Other): All adult patients with kidney failure referred to a department of renal medicine at one of the four hospitals from the 1st of October 2016 to the 31st of May 2018 were offered the intervention and invited to participate in the study. The inclusion criterion was an estimated glomerular filtration rate below 20 ml/min and based on a clinical judgement made by the contact doctor and/or the contact nurse about the decline in the Estimated glomerular filtration rate to continue. Exclusion criteria were patients who had decided on conservative management, patients with a living donor and a set date for transplantation and patients not able to participate in the intervention due to cognitive impairment. The use of an interpreter was not an exclusion criterion.
  Interventions: Other: SDM-DC

INTERVENTIONS:
Other: SDM-DC — The SDM-DC intervention is designed for patients with kidney failure who must make a decision regarding type of dialysis: haemodialysis or peritoneal dialysis. SDM-DC consists of patient and his or her relative(s) being given a patient decision aid called 'Dialysis choice' and booked for meetings with a dialysis coordinator. There were optional videos describing other patients' experiences making this decision. The dialysis coordinators were trained in the why, what and how in relation to SDM-DC and to deliver the intervention by tailoring to patients' needs and using three different communication skills: mirroring, active listening and value clarification.
  Other Names: Shared decision-making and dialysis choice

SUMMARY:
The SDM-DC intervention is designed for patients with kidney failure who must make a decision regarding type of dialysis: haemodialysis or peritoneal dialysis. SDM-DC consists of patient and his or her relative(s) being given a patient decision aid called 'Dialysis choice' and booked for meetings with a dialysis coordinator.

DETAILED DESCRIPTION:
The dialysis coordinators were trained in the why, what and how in relation to SDM-DC and to deliver the intervention by tailoring to patients' needs and using three different communication skills: mirroring, active listening and value clarification. The patient decision aid was designed to be utilised during and between the SDM-DC meetings. The patient decision aid is in paper format and consists of a set of tools: a decision map, an overview of uremic symptoms, an overview of options, and the Ottawa Personal Decision Guide. More specifically, the patient decision aid makes explicit the dialysis decision, describes options, benefits and harms using the best available evidence, and intends to help patients clarify their values by indicating the importance of the benefits and harms out of scale from (0) to (5). Four videos with personal stories were available to be shown and discussed at the meetings if the patient preferred to see the reason why another patient has chosen a specific option. Each video showed one option with a patient telling why he/she chose that option, and how he/she weighed the advantages and disadvantages.

ELIGIBILITY:
Inclusion Criteria:

* Estimated glomerular filtration rate below 20 ml/min
* A clinical judgement made by the contact nurse and the contact physician

Exclusion Criteria:

* Conservative care
* A set date for a transplantation with a living donor
* Not able to participate due to cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Patients experiences of a shared decision-making process | 14 days after interventions
  Shared decision-making questionnaire was used to measure patients' perception of shared decision-making in the clinical encounter. It consists of nine statements to be rated on a six-point scale from 'completely disagree' (0) to 'completely agree' (5) The quality of the decision-making process was calculated as the mean score for each item in the SDM-Q9. To provide a total score of the SDM-Q9 a sum of all items was calculated and standardized on a scale on 0-100.
Knowledge, readiness for decision-making and decision quality | 14 days after interventions
  Decision Quality Measurement was used to measure the quality of the decision. The questionnaire consists of six knowledge statements and six readiness statements. All items on the questionnaire were rated as yes, no or unsure. It also consists of two open questions. A total knowledge and readiness score was calculated and standardized out of 100. Open questions were analysed using descriptive qualitative analysis and reported based on most common to least common comments. We decided that for a home-based treatment and choosing 'Treatment at home' in the preference question or deciding for a hospital-based treatment and not choosing 'Treatment at home' in the preference question were considered as concordant choices. Decision quality was defined as a knowledge score >66% on the knowledge score and combined with the concordance score.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanette Finderup, Master, Principal Investigator — Aarhus University Hospital

IPD SHARING:
Plan to Share IPD: No
The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request. But restrictions apply to the availability of these data, which were used under license for the current study, and so are not publicly available.

REFERENCES:
- [Derived] Finderup J, Lomborg K, Jensen JD, Stacey D. Choice of dialysis modality: patients' experiences and quality of decision after shared decision-making. BMC Nephrol. 2020 Aug 5;21(1):330. doi: 10.1186/s12882-020-01956-w. PMID 32758177